CLINICAL TRIAL: NCT01234038
Title: A Phase 1b/2 Study of Carboplatin-Paclitaxel, With or Without ISIS 183750 (an eIF4E Inhibitor), in Patients With Stage IV Non-Small Cell Lung Cancer
Brief Title: Safety and Tolerability Study of ISIS EIF4E Rx in Combination With Carboplatin and Paclitaxel
Acronym: NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 183750-CS4
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 Cohort 1 (Experimental)
  Interventions: Drug: ISIS EIF4E Rx; Drug: Paclitaxel; Drug: Carboplatin
- Part 1 Cohort 2 (Experimental)
  Interventions: Drug: ISIS EIF4E Rx; Drug: Paclitaxel; Drug: Carboplatin
- Part 2 Arm A (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Part 2 Arm B (Experimental)
  Interventions: Drug: ISIS EIF4E Rx; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: ISIS EIF4E Rx — 800 mg ISIS EIF4E Rx administered as a 3-hour intravenous infusion on Days 1, 8 and 15 of each 21 day cycle
  Arms: Part 1 Cohort 1
Drug: ISIS EIF4E Rx — 1000 mg ISIS EIF4E Rx administered as a 3-hour intravenous infusion on Days 1, 8 and 15 of each 21 day cycle
  Arms: Part 1 Cohort 2
Drug: ISIS EIF4E Rx — (Dose identified in Part 1)ISIS EIF4E Rx administered as a 3-hour intravenous infusion on Days 1, 8, and 15 of each 21 day cycle
  Arms: Part 2 Arm B
Drug: Paclitaxel — 200 mg/m2 administered as a 3-hour intravenous infusion on Day 1 of each 21 day cycle
Drug: Carboplatin — AUC 6.0 mg/mL/min administered as a 1-hour intravenous infusion on Day 1 of each 21 day cycle

SUMMARY:
The purpose of this study is to examine the overall survival of patients with Stage IV non-small cell lung cancer (NSCLC) treated with ISIS EIF4E Rx in combination with carboplatin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age >/= 18 years
* Histologically or cytologically confirmed diagnosis of NSCLC
* Stage IV disease (including patients with pleural effusion who were previously classified as Stage IIIB)
* All of the following if patient has had prior radiation therapy:

  1. Lesion(s) used for determination of response were not previously irradiated or have increased in size since the completion of radiotherapy
  2. The patient has recovered from any acute effects of the radiotherapy
  3. Radiotherapy was completed at least 4 weeks prior to Screening
* Part 1: Have at least non-measurable evaluable disease (e.g., lesions which are smaller than the minimum size required for measurability; other non-measurable lesions such as bone metastases, malignant pleural effusion)
* Part 2: Have measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension
* Performance status of 0 or 1 on the ECOG Performance Status Scale
* Have an estimated life expectancy of at least 12 weeks
* Adequate organ function within 14 days prior to first study dose (ISIS EIF4E Rx or carboplatin/paclitaxel, whichever occurs first) as defined by:

  1. Absolute neutrophil count (ANC) >/= 1.5 x 109/L
  2. Platelet count >/= 100 x 109/L
  3. Hemoglobin >/=9 g/dL (>/= 5.6 mmol/L). Patients may receive packed RBC transfusion to achieve this level at the discretion of the investigator.
  4. Total bilirubin < 1.5 x upper limit of normal (ULN) unless elevated secondary to conditions such as Gilbert's Disease
  5. Aspartate aminotransferase (AST) < 3 x ULN (< 5 x ULN in the presence of hepatic metastases)
  6. Alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN in the presence of hepatic metastases)
  7. Alkaline phosphatase < 3.0 x ULN
  8. Calculated creatinine clearance >/= 60 mL/min per Cockcroft and Gault formula
* Satisfy one of the following:

  1. Females: non-pregnant and non-lactating; surgically sterile, post-menopausal, or patient or partner compliant with a reliable contraceptive regimen, as determined by Investigator, for 4 weeks prior to Screening. Patients of reproductive potential must test negative for pregnancy at Screen and must agree to use a reliable method of birth control during the study and for the 10 weeks following the last dose of ISIS EIF4E Rx.
  2. Males: surgically sterile or patient or partner must agree to use a reliable contraceptive method, as determined by the Investigator during the study and for the 10 weeks following the last dose of ISIS EIF4E Rx.
* For Part 1: have discontinued all prior chemotherapies, biological therapies, and other investigational therapies for cancer for at least 4 weeks (6 weeks for mitomycin-C or nitrosoureas) prior to study treatment and recovered from the acute effects of therapy.

Exclusion Criteria:

* Part 1: More than 2 prior chemotherapy or biological therapy regimens (approved or experimental) for NSCLC, not counting adjuvant and neoadjuvant treatment. A regimen is defined as two or more consecutive cycles of treatment.
* Part 2: Any prior chemotherapy or biological therapy (approved or experimental) for NSCLC including adjuvant and neoadjuvant treatments
* Treatment with another investigational drug, biological agent, or device within 4 weeks (6 weeks for biological agents) before Screening or 5 half-lives of study agent, whichever is longer
* Patients with treated or untreated parenchymal brain metastases or leptomeningeal disease. Brain imaging is required for symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients.
* Patients with known pericardial effusion
* Have active infection or serious concomitant systemic disorder (for example, heart failure) incompatible with the study (at the discretion of the Investigator)
* Presence or history of malignancy other than NSCLC, carcinoma in situ of the cervix, or non-melanoma skin cancer. In the case of other malignancies, patients may be considered for participation if the prior malignancies were diagnosed and definitively treated at least five years previously with no subsequent evidence of recurrence.
* Presence of an underlying disease state associated with active bleeding
* Ongoing therapy with oral or parenteral anticoagulants (e.g., heparin, warfarin/coumadin). Low-dose anticoagulants for maintenance of catheter patency and low dose aspirin (≤ 325 mg/day) and nonsteroidal anti-inflammatory agents are not exclusionary.
* Concurrent treatment with other anticancer drugs
* Pre-existing peripheral neuropathy >/=Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE) Grade 2
* Known history of HIV, HCV, or chronic HBV infection
* Previous treatment with a therapeutic antisense oligonucleotide or siRNA
* Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device
* Have any other medical conditions that in the opinion of the Investigator, would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | At the end of each 21 day cycle

CONTACTS AND LOCATIONS:
Locations (29):
- United States (10):
  - Achieve Clinical Research, Birmingham, Alabama
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Little Rock Cancer Clinic, Little Rock, Arkansas
  - Kenmar Research Institute, Los Angeles, California
  - Joliet Hematology Oncology Associates, Joliet, Illinois
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - Jewish Hospital & St. Mary's Healthcare, Louisville, Kentucky
  - Gabrail Cancer Center, Canton, Ohio
  - Cancer Therapy and Research Center, University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Hungary (5):
  - Koranyi National Institute of TBC and Pulmonology, Budapest
  - Semmelweis University Faculty of Medicine, Budapest
  - University of Debrecen, Medical and Health Science Center, Debrecen
  - Hospital for Thoracic Diseases of Csongrad County Local Governmental, Deszk
  - Bekes Country Pandy Kalman Hospital, Gyula
- Poland (5):
  - K. Dluski Provincial Specialist Hospital, Bialystok
  - Independent Public Teaching Hospital No. 4 In Lublin, Lublin
  - Idependent Public Tuberculosis an Lung Diseases Facilities, Olsztyn
  - Specialist Tuberculosis and Lung Diseases Hospitals, Rzeszów
  - Alojzy Pawelec Provincial Hospital of Lung Diseases, Wodzisław Śląski
- Russia (9):
  - State Medical Institution: Arkhangelsk Regional Clinical Oncology Center, Chemotherapy department, Arkhangelsk
  - State Therapeutical and Prophylactic Institution: Chelyabinsk Regional Clinical Oncology Center, Chemotherapy Department, Chelyabinsk
  - State Healthcare Institution: Ivanovo Regional Oncology Center, Chemotherapy Department, Ivanovo
  - Non-State Medical Institution: Central Clinical Hospital #2 n.a. N.A. Semashko under OJSC Russian Railways, Chemotherapy Dept., Moscow
  - State Healthcare Institution: Leningrad Regional Clinical Hospital, Thoracic Surgery Department, Saint Petersburg
  - St. Petersburg State Healthcare Institution: "City Clinical Oncology Center", Saint Petersburg
  - State Higher Educational Institution: St. Petersburg State Medica University n.a.I.P. Pavlov under the Federal Agency for Healthcare and Social Development, Pulmonology Research Institute, Saint Petersburg
  - State Institution: Samara Regional Clinical Oncology Center, Chemotherapy Department, Samara
  - State Budget Healthcare Institution: Sverdlovsk Regional Oncology Center, Radiotherapy Department, Yekaterinburg